CLINICAL TRIAL: NCT00606502
Title: A Randomized, Phase 2b, Multi-center Study of Pralatrexate Versus Erlotinib in Patients With Stage IIIB/IV Non-small Cell Lung Cancer After Failure of at Least 1 Prior Platinum-based Treatment
Brief Title: Study of Pralatrexate vs. Erlotinib for Non-Small Cell Lung Cancer After at Least 1 Prior Platinum-based Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDX-012; 2007-004673-26 (EudraCT Number)
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Results first posted 2011-01-20 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Stage IIIB/IV non-small cell lung cancer; Non-small cell lung cancer; NSCLC; Lung Cancer; Pralatrexate; Erlotinib; Tarceva; PDX; Smoking; Smoker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Smoking | interventions — 10-propargyl-10-deazaaminopterin; Erlotinib Hydrochloride; Vitamin B 12; Folic Acid

ARMS (2):
- Pralatrexate (Experimental): Intravenous (IV) push administration over 3-5 minutes into a patent IV line containing normal saline (0.9% sodium chloride).
  Interventions: Drug: Pralatrexate; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid
- Erlotinib (Active Comparator): 150 mg orally in tablet form
  Administered daily 1 hour before or 2 hours after ingestion of food until criteria for discontinuation per the protocol are met.
  Interventions: Drug: Erlotinib; Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid

INTERVENTIONS:
Drug: Pralatrexate — Intravenous (IV) push administration over 3-5 minutes into a patent IV line containing normal saline (0.9% sodium chloride).
  Initial dose: 230 mg/m2, increased to 270 mg/m2 if patient does not have specific adverse events (AEs) as per the protocol after receipt of 2 consecutive doses 2 weeks apart. Reductions allowed in 40 mg/m2 decrements to 190 mg/m2 per the protocol defined dose modifications.
  Protocol amended dose: 190 mg/m2, then 230 mg/m2 if patient does not have specific AEs per the protocol after receipt of 2 consecutive doses 2 weeks apart. Reductions allowed in 40 mg/2 decrements to 150 mg/m2 per the protocol defined dose modifications.
  Administered on days 1 and 15 of a 4-week cycle (every 2 weeks) until criteria for discontinuation per the protocol are met.
  Other Names: FOLOTYN; PDX; (RS)-10-propargyl-10-deazaaminopterin
  Arms: Pralatrexate
Drug: Erlotinib — 150 mg orally in tablet form
  Administered daily 1 hour before or 2 hours after ingestion of food until criteria for discontinuation per the protocol are met.
  Other Names: Tarceva®; Erlotinib hydrochloride
  Arms: Erlotinib
Dietary Supplement: Vitamin B12 — 1 mg intramuscular injection
  Administered within 10 weeks of randomization, every 8-10 weeks throughout the study and for at least 30 days after last dose of study treatment.
  Other Names: Cyanocobalamin
Dietary Supplement: Folic Acid — 1-1.25 mg orally
  Administered daily for at least 7 days prior to randomization, throughout the study and for at least 30 days after last dose of study treatment.
  Other Names: Vitamin B9; Folate; Folacin

SUMMARY:
The purpose of this clinical study is to determine the effectiveness (ability to provide beneficial treatment of the disease) and safety of pralatrexate compared to erlotinib when given to non-small cell lung cancer (NSCLC) patients who are current or former cigarette smokers and who have received at least 1 prior treatment with a platinum drug (cisplatin or carboplatin)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Stage IIIB/ IV non-small cell lung cancer (NSCLC).
* Relapsed after treatment with 1 or 2 prior chemotherapy regimens, including at least 1 platinum-based treatment. Patients may have received pemetrexed as 1 of the prior therapies. Patients may not have received investigational therapy as their only prior therapy.
* Recovered from the toxic effects of prior therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Smoked ≥ 100 cigarettes in their lifetime, whether a former or current cigarette smoker.
* Adequate blood, liver and kidney function as defined by laboratory values.
* Received 1-1.25 mg daily oral folic acid for at least 7 days prior to randomization and 1 mg intramuscular injection of vitamin B12 within 10 weeks prior to randomization.
* Women of childbearing potential must use medically acceptable birth control and have a negative serum pregnancy test within 14 days prior to randomization. Patients who are postmenopausal for at least 1 year (> 12 months since last menses) or are surgically sterilized do not require this test.
* Men who are not surgically sterile must use medically safe and effective birth control from the time of study randomization, and agree to continue practicing until at least 90 days after the last administration of study treatment.
* Accessible for repeat dosing and follow-up.
* Give written informed consent.

Exclusion Criteria:

* Active concurrent primary malignancy (except non-melanoma skin cancer or in situ carcinoma of the cervix). If there is a history of prior malignancy, the patient must be disease-free for ≥ 5 years. Patients with other prior malignancies less than 5 years before study entry may still be enrolled if they have received treatment resulting in complete resolution of the cancer and currently have no evidence of active or recurrent disease.
* Use of investigational drugs, biologics, or devices within 4 weeks prior to randomization.
* Previous exposure to pralatrexate or erlotinib.
* Women who are pregnant or breastfeeding.
* Congestive Heart Failure Class III/IV according to New York Heart Association (NYHA) Functional Classification.
* Uncontrolled hypertension.
* Human immunodeficiency virus (HIV)-positive diagnosis with a CD4 count of <100 mm3 or detectable viral load within the past 3 months, and is receiving combination anti-retroviral therapy.
* Symptomatic central nervous system metastases or lesions for which treatment is required.
* Major surgery within 2 weeks of study randomization.
* Receipt of any conventional systemic chemotherapy within 4 weeks (6 weeks for nitrosoureas, mitomycin C), or radiation therapy (RT) within 2 weeks, prior to randomization.
* Active infection or any serious underlying medical condition, which would impair the ability of the patient to receive protocol treatment.
* Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent or limit study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06-24 (Actual); Study Completion 2010-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garry Weems, PharmD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (47):
- United States (15):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Sharp Memorial Hospital, San Diego, California
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Donald Berdeaux, Great Falls, Montana
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Hematology and Oncology Associates South Jersey, Mount Holly, New Jersey
  - New York Oncology Hematology-Oncology Associates, P.C., Latham, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New Bern Cancer Care, New Bern, North Carolina
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Baptist Regional Cancer Center, Knoxville, Tennessee
  - Cancer Therapy and Research Center, San Antonio, Texas
  - Providence Everett Medical Center, Everett, Washington
- Argentina (6):
  - Policlinica Privada - Instituto de Medicina Nuclear, Bahía Blanca, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires, Cuidad de Buenos Aires
  - Hospital Britanico, Capital Federal
  - Centro Oncologico Rosario, Rosario
  - CAIPO (Centero Para la Atencion Integral del Paciente Oncologico), San Miguel de Tucumán
  - ISIS Clinica Especializada, Santa Fe
- Brazil (6):
  - Associação Hospital de Caridade de Ijuí, Ijuí, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Clinionco - Clínica de Oncologia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital do Câncer de Barretos, Barretos, São Paulo
  - Biocancer S.A., Belo Horizonte
  - Instituto do Cancer - Arnaldo Vieira de Carvalho, São Paulo
- Czechia (6):
  - Masarykuv onkologicky ustav, Brno
  - Palacký University Medical School and Teaching Hospital, Olomouc
  - Vitkovicka nemocnice, a. s., Ostrava
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Na Homolce, Prague
  - Fakultni nemocnice na Bulovce, Prague
- Hungary (6):
  - National Koranyi TBC and Pulmonology Institute, Budapest, Pest County
  - Jósa András Teaching Hospital, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Vas County Markusovszky Hospital, Szombathely, Vas County
  - Zala County Hospital, Zalaegerszeg, Zala County
  - Matrai Allami Gyogyintezet, Mátraháza
  - Komarom-Esztergom Megyei Onkorm. Szent Borbala Korhaza, Tatabánya
- India (8):
  - MNJ Radium Hospital and Radium Institute of Oncology and Regional Cancer Centre, Hyderabaad, Andhra Pradesh
  - Indo American Cancer Institute and Research Center, Hyderabad, Andhra Pradesh
  - Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - Regional Cancer Center, Trivandrum, Kerala
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Jehangir Clinical Development Centre Pvt Ltd, Pune, Mahara
  - B.P. Poddar Cancer Institute, Kolkata, West Bengal
  - Dharmashila Cancer Hospital & Research Centre, New Delhi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between January 2008 and June 2009 across 43 study sites in 6 countries.
Groups:
- Pralatrexate: 190 or 230 mg/m2 starting dose with increases or decreases to 150 to 270 mg/m2 per protocol, administered as an IV push over 3-5 minutes on days 1 and 15 of a 4-week cycle (ie, every 2 weeks)
- Erlotinib: 150 mg tablet taken orally daily
Period: Randomization
Arm/Group | Pralatrexate | Erlotinib
Started | 100 | 101
Completed | 97 | 101
Not Completed | 3 | 0
Not completed — Randomized but not treated | 3 | 0
Period: Treatment
Arm/Group | Pralatrexate | Erlotinib
Started | 97 | 101
Completed | 97 | 98
Not Completed | 0 | 3
Not completed — Treatment ongoing at time of data cutoff | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pralatrexate | Erlotinib | Total
Number analyzed (Participants) | 100 | 101 | 201
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 58 | 60 | 118
  >=65 years | 42 | 41 | 83
Age, Continuous [Median (Standard Deviation); unit: years] | 63.0 (9.0) | 62.0 (9.1) | 63.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 69 | 68 | 137
Region of Enrollment [Number; unit: participants]
  United States | 31 | 37 | 68
  Czech Republic | 17 | 20 | 37
  Hungary | 17 | 15 | 32
  India | 11 | 12 | 23
  Brazil | 13 | 9 | 22
  Argentina | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) of Patients Receiving Pralatrexate vs. Erlotinib
Description: OS was defined as the length of time from randomization until death due to any cause. Patients who were alive at the time of the data cut-off date were censored at the last contact date.
Time Frame: Assessed from date of randomization no less frequently than every 16 weeks for up to 2 years after randomization.
Measure: Median (95% Confidence Interval); unit: Months Survival
Arm/Group | Pralatrexate | Erlotinib
Number analyzed (Participants) | 100 | 101
Months Survival | 6.7 [5.3 to 9.0] | 7.0 [3.9 to 7.9]
Statistical Analysis 1: Comparison: Pralatrexate vs Erlotinib; Test type: Superiority or Other; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.61 to 1.14]

2. Secondary Outcome: Response Rate (RR) to Treatment of Patients Receiving Pralatrexate vs. Erlotinib
Description: Number of patients whose tumors responded to Pralatrexate or Erlotinib, using the Response Criteria in Solid Tumors (RECIST).
Time Frame: Assessed every 8 weeks for the first 24 weeks, then every 16 weeks for up to 2 years or until PD or start of subsequent treatment.
Population: Based on all treated patients with measurable disease at baseline. Patients who were declared unevaluable for response were considered nonresponders and were included in the calculation of response rate. Patients were unevaluable if they were off-treatment prior to first response assessment, never received treatment or had unconfirmed responses.
Measure: Number; unit: Participants
Arm/Group | Pralatrexate | Erlotinib
Number analyzed (Participants) | 97 | 98
Participants
  Complete + Partial Response | 2 | 7
  Complete Response (CR) | 0 | 1
  Partial Response (PR) | 2 | 6
  Stable Disease (SD) | 33 | 35
  Progressive Disease (PD) | 29 | 36
  Disease Control (CR+PR+SD) | 35 | 42
  Unable to Evaluate | 2 | 0
  Missing (off or no treatment, not confirmed) | 31 | 20

3. Secondary Outcome: Progression-free Survival (PFS) of Patients Receiving Pralatrexate vs. Erlotinib
Description: PFS was calculated as the number of days from randomization to the date of radiological evidence of PD or death due to any cause.
Time Frame: as for outcome 2
Population: Patients who were alive without a disease response assessment of PD as of the data cut-off date were censored at the last disease assessment date or the date of randomization, whichever was later. Patients with no response assessments after baseline were censored at date of randomization resulting in a duration of PFS of 1 day.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pralatrexate | Erlotinib
Number analyzed (Participants) | 100 | 101
months | 3.4 [2.1 to 4.7] | 2.8 [2.1 to 3.7]

4. Secondary Outcome: Adverse Events of Patients Receiving Pralatrexate vs. Erlotinib
Time Frame: Assessed every 2 weeks while on treatment through safety follow-up visit (35 +/-5 days post-last dose) or early termination visit (at time of withdrawal).
Population: Adverse Events (AEs) and Serious AEs (SAEs) are presented regardless of causality for patients who received at least one dose of Pralatrexate or Erlotinib. Events were graded by the investigator using the NCI CTCAE Scale (version 3.0) which provides a grading scale for each AE term.
  Grade 3 = Severe
  Grade 4 = Life-threatening or disabling
Measure: Number; unit: Treated Participants
Arm/Group | Pralatrexate | Erlotinib
Number analyzed (Participants) | 97 | 101
Treated Participants
  At least one AE | 75 | 77
  Grade 3 AEs | 25 | 18
  Grade 4 AEs | 5 | 0
  At least one SAE | 14 | 2

ADVERSE EVENTS:
Time Frame: Assessed every 2 weeks while on treatment through safety follow-up visit (35 +/-5 days post-last dose) or early termination visit (at time of withdrawal).
Description: Events reported for all patients who received at least one dose of Pralatrexate or Erlotinib.
Arm/Group | Pralatrexate | Erlotinib
Serious Adverse Events (participants affected / at risk) | 31/97 | 32/101
Other Adverse Events (participants affected / at risk) | 91/97 | 94/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pralatrexate (N=97) | Erlotinib (N=101)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 1
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
stomatitis (Gastrointestinal disorders) | 9 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 3
diarrhoea (Gastrointestinal disorders) | 1 | 1
gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
vomiting (Gastrointestinal disorders) | 0 | 2
anal inflammation (Gastrointestinal disorders) | 1 | 0
dysphagia (Gastrointestinal disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 0 | 1
sepsis (Infections and infestations) | 3 | 3
pneumonia (Infections and infestations) | 2 | 3
respiratory tract infection (Infections and infestations) | 1 | 1
chest wall abscess (Infections and infestations) | 0 | 1
infection (Infections and infestations) | 1 | 0
influenza (Infections and infestations) | 1 | 0
pulmonary sepsis (Infections and infestations) | 0 | 1
septic shock (Infections and infestations) | 1 | 0
urosepsis (Infections and infestations) | 0 | 1
pyrexia (General disorders) | 2 | 4
asthenia (General disorders) | 0 | 1
fatigue (General disorders) | 1 | 0
multimorbidity (General disorders) | 1 | 0
non-cardiac chest pain (General disorders) | 0 | 1
sudden death (General disorders) | 1 | 0
dehydration (Metabolism and nutrition disorders) | 1 | 4
anorexia (Metabolism and nutrition disorders) | 0 | 1
hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
leukopenia (Blood and lymphatic system disorders) | 3 | 0
anaemia (Blood and lymphatic system disorders) | 2 | 0
neutropenia (Blood and lymphatic system disorders) | 1 | 0
pancytopenia (Blood and lymphatic system disorders) | 1 | 0
pericardial effusion (Cardiac disorders) | 1 | 2
atrial fibrillation (Cardiac disorders) | 1 | 1
cardio-respiratory arrest (Cardiac disorders) | 1 | 1
convulsion (Nervous system disorders) | 1 | 3
cerebral infarction (Nervous system disorders) | 0 | 1
headache (Nervous system disorders) | 1 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
arterial thrombosis (Vascular disorders) | 0 | 1
deep vein thrombosis (Vascular disorders) | 1 | 0
hypotension (Vascular disorders) | 1 | 0
bile duct obstruction (Hepatobiliary disorders) | 1 | 0
hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
femur fracture (Injury, poisoning and procedural complications) | 1 | 1
cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
confusional state (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pralatrexate (N=97) | Erlotinib (N=101)
stomatitis (Gastrointestinal disorders) | 62 | 4
diarrhoea (Gastrointestinal disorders) | 15 | 32
nausea (Gastrointestinal disorders) | 12 | 17
vomiting (Gastrointestinal disorders) | 10 | 10
constipation (Gastrointestinal disorders) | 3 | 8
dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 28
rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 21
dry skin (Skin and subcutaneous tissue disorders) | 2 | 9
fatigue (General disorders) | 25 | 16
asthenia (General disorders) | 15 | 8
oedema peripheral (General disorders) | 5 | 7
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 22
cough (Respiratory, thoracic and mediastinal disorders) | 11 | 17
anorexia (Metabolism and nutrition disorders) | 16 | 19
hypokalaemia (Metabolism and nutrition disorders) | 5 | 8
back pain (Musculoskeletal and connective tissue disorders) | 3 | 10
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 9
anaemia (Blood and lymphatic system disorders) | 20 | 12
thrombocytopenia (Blood and lymphatic system disorders) | 12 | 1
bronchitis (Infections and infestations) | 5 | 8
weight decreased (Investigations) | 8 | 10
conjunctivitis (Eye disorders) | 6 | 5

LIMITATIONS AND CAVEATS:
The date of the CRF database cut-off for patients (no further case report form or query data entry) was 24 Jun 2010. As of the CRF data cut-off date, 3 patients, remained on therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Allos agreements with investigators (PIs) may vary. The PI may publish/make public data from the study after the earlier of publication by Allos or 24 months after database lock. Allos is allowed 60 days to review and comment on the communication prior to public release. Allos can request removal of confidential information (other than study results).